CLINICAL TRIAL: NCT07072728
Title: A Phase 2b Double-blind, Randomized, Low-dose Comparator-controlled Clinical Trial to Assess the Efficacy and Safety of PEX010 in Psilocybin-assisted Psychotherapy for the Treatment of Adjustment Disorder Associated With Cancer.
Brief Title: Psilocybin-Assisted Psychotherapy in Cancer Patients With Adjustment Disorder
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Psyence Australia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PSY-01
Record Dates: First submitted 2025-02-12; First posted 2025-07-18 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Adjustment Disorder; Adjustment Disorder With Anxious Mood; Cancer; Cancer Cachexia; Cancer of Endometrium; Cancer of Kidney; Cancer of Prostate; Cancer of the Breast; Cancer of Stomach; Cancer Melanoma Skin; Cancer Pancreas
Keywords: Cancer; Adjustment Disorder; Existential Distress; Psilocybin; Psilocin
MeSH Terms: conditions — Adjustment Disorders; Neoplasms; Endometrial Neoplasms; Kidney Neoplasms; Prostatic Neoplasms; Breast Neoplasms; Stomach Neoplasms; Melanoma; Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants will be centrally randomized 1:1:1 to a treatment group.
  * Group 1: 25 mg PEX010;
  * Group 2: 10 mg PEX010;
  * Group 3: 1 mg PEX010 (low-dose comparator).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1: 25 mg PEX010 Psilocybin Capsules (Active Comparator): Participants in Group 1 will receive a single dose of 25 mg PEX010 psilocybin capsules under medical supervision on Day 14. Non-responders at Week 10, who continue to meet eligibility criteria, may receive a second cycle of psilocybin-assisted psychotherapy (PAP) at the same 25 mg dose. A maximum of two PAP cycles may be administered.
  Interventions: Drug: Psilocybin therapy
- Group 2: 10 mg PEX010 Psilocybin Capsules (Active Comparator): Participants in Group 2 will receive a single dose of 10mg PEX010 psilocybin capsules under medical supervision on Day 14. Non-responders at Week 10, who continue to meet eligibility criteria, may receive a second cycle of psilocybin-assisted psychotherapy (PAP) at the 25 mg dose. A maximum of two PAP cycles may be administered.
  Interventions: Drug: Psilocybin therapy
- Group 3: 1 mg PEX010 (low-dose comparator) (Placebo Comparator): Participants in Group 3 will receive a single dose of 1mg PEX010 psilocybin capsules under medical supervision on Day 14. Non-responders at Week 10, who continue to meet eligibility criteria, may receive a second cycle of psilocybin-assisted psychotherapy (PAP) at the same 25 mg dose. A maximum of two PAP cycles may be administered.
  Interventions: Drug: Psilocybin therapy

INTERVENTIONS:
Drug: Psilocybin therapy — Following a screening period, eligible participants will undergo one cycle of psilocybin-assisted psychotherapy (PAP). Non-responders at Week 10 who continue to meet eligibility criteria will be offered a second PAP cycle at the 25 mg PEX010 dose. A maximum of two PAP cycles may be given. Long-term follow-up will include a visit at Month 3 following the final PAP cycle.

SUMMARY:
This study is assessing the efficacy and safety of PEX010 in psilocybin-assisted psychotherapy for the treatment of adjustment disorder due to cancer diagnosis.

Who is it for? This study is for people who are aged between 18 and 80 years old and suffer from anxiety after adjusting to an acutely stressful event of their cancer diagnosis. This is called adjustment disorder.

Study details Participants in this study will be randomly allocated by chance (similar to flipping a coin) to one of three groups: a 25mg PEX010 dose group, a 10 mg PEX010 dose group or a 1mg PEX010 dose group. Participants will be allocated a dose that will be administered during their psilocybin-assisted psychotherapy (PAP) dosing session. The PAP dosing session will run approximately 8 hours, with PEX010 administered at Day 14 (dosing day).

At Week 10, non-responders that continue to meet the study eligibility criteria may commence an additional PAP cycle (at 25 mg PEX010). A maximum of 2 PAP cycles may be administered. Long term follow up will comprise of a study visit at 3 months post Week 10 (of the final cycle) to assess safety and tolerability of PEX010.

It is hoped that this research will develop important scientific knowledge that could contribute to the development of a potential new treatment for anxiety and depression after adjusting to an acutely stressful event such as a cancer diagnosis.

DETAILED DESCRIPTION:
This is a randomized, double-blind, low-dose comparator-controlled Phase IIb study to investigate the efficacy and safety of PAP with 25 mg, 10 mg and 1 mg [low-dose comparator) PEX010, for the treatment of adjustment disorder symptoms in participants diagnosed with cancer. The referring oncologist will indicate that the participant is physically capable of undergoing psychedelic encounter and is likely to have a minimum life expectancy of 6 months.

At least 87 adult participants (age 18 to 80 at screening) with a diagnosis of AjD due to cancer diagnosis will be enrolled in this study. Participants will be randomly assigned with a ratio of 1:1:1 to receive Psilocybin-Assisted Psychotherapy (PAP) with either 25 mg, 10 mg or 1 mg PEX010. Both the site staff treating participants and the participants themselves will be blinded to the treatments being administered.

The study consists of a combination of clinic visits and telehealth phone calls to support this vulnerable participant population. The clinic will have experience with conducting PAP. All study visits be carried out by suitably qualified individuals and wherever possible, the same therapist will meet with study participants for in-person and telehealth appointments. Participants will undertake a screening visit between Day -28 and Day -2 to determine eligibility to participate in the study. Those participants that meet the eligibility criteria will attend the study site on Day 1 when continued eligibility will be assessed and baseline assessments performed.

Participants must complete three preparation sessions with the therapist prior to dosing session. Two of these sessions can be completed remotely via telehealth and have flexible timing, provided there is at least one day between each session. One preparation session must be done in person in the dosing room, ideally during a site visit on Day 13. Additionally, at least one preparation session must include the sitter or secondary therapist. The primary therapist has the discretion to include the sitter or secondary therapist in more preparation or integration sessions based on their assessment.

The clinic site visits will comprise Day 1, Day 13 (day prior dosing session), Day 14 (dosing session), Day 15 (integration session) and Day 70/Week 10 (follow-up) post-randomization. There will be ± 3 days for a dosing session allowed. Subsequently, all relevant visits will be adjusted accordingly. In addition, participants will be required to attend following telehealth appointments:

* Two telehealth appointments for preparatory sessions within 2 weeks prior to dosing session.
* One telehealth appointment for integration therapy session in the two weeks following the dosing session.
* Follow up telehealth appointments on Day 28 (Week 4), Day 42 (Week 6).
* Final study follow-up telehealth appointment at 3 months post the Day 70 (Week 10) visit of the final PAP cycle for final safety assessments.

Non responders (for criteria see Section 5.5.2) at Day 70 (Week 10) that continue to meet the study eligibility criteria, may commence an additional PAP cycle (at 25 mg PEX010). These participants will repeat the schedule described above, including the visit the day prior to dosing session, the actual dosing session, and the integration sessions. A maximum of 2 PAP cycles may be administered.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for study entry participants must satisfy all of the following criteria:

1. Screening AjD diagnosis (ICD-11), as defined by an ADNM-20 score ≥ 47.5, a score of ≥ 4 on the Distress Thermometer.
2. Screening HAM-A Score ≥18 (moderate anxiety).
3. Adults aged 18 to 80 years (inclusive) at screening.
4. Diagnosed with cancer (exempting those cancers listed in the exclusion criteria) and a minimum life-expectancy of 6 months in the opinion of the treating physician, with performance status of 0-2 on the Eastern Cooperative Oncology Group (ECOG) scale performed at screening.
5. Agrees not to commence any new psychiatric medications or psychotherapies from Screening to Week 10.
6. Able to communicate well and follow study procedures, judged as sufficiently competent with the English language by the investigator, able to build adequate rapport with study staff.
7. Judged to be of low suicide risk based on Sheehan-Suicide Tracking Scale (S-STS) and the opinion of a research team psychiatrist.
8. Be medically suitable in the opinion of the investigator as determined by screening for medical problems via a personal interview, a medical questionnaire, a physical examination, an electrocardiogram (ECG), and blood tests.
9. Have access to a device that is compatible to use the digital technology, i.e smart-phone device tablet.
10. Agree not to take any sedating medications for a minimum of 12 hours before the dosing session including benzodiazepines, zopiclone, eszopiclone, zaleplon and zolpidem. Medications for cancer-related pain are permitted.
11. Must be willing and able to refrain from smoking throughout the duration of the dosing session. Nicotine replacement therapies may be permitted with the agreement of the medical monitor.
12. Agree that for 1 week before the psilocybin dosing session, participants will refrain from taking any illegal drugs or non-prescription medication (including cannabis, or CBD or THC containing products), nutritional supplement, or herbal supplement except when approved by the study investigators. Additionally, agree not to take any form of psilocybin outside of the study, including microdosing, from baseline through Day 70/Week 10 (Visit 11).
13. Participants taking any other medication that is not explicitly detailed as an excluded medication will be discussed with the investigator and medical monitor as appropriate. Decisions on inclusion will be based on clinical judgement and with sufficient justification provided.

Exclusion Criteria

Participants will be excluded from the study if one or more of the following criteria are applicable:

Psychiatric Exclusion Criteria:

1. Current Major Depressive Disorder MDD (or within 12 months of Screening) deemed independent from the cancer diagnosis, current or past diagnosis of schizophrenia, psychotic disorder, unless this was resulting from a medical condition (e.g. lupus or malaria etc.), bipolar disorder I and II, delusional disorder, paranoid personality disorder, schizoaffective disorder, borderline personality disorder, anti-social personality disorder or judged to be incompatible with establishment of rapport or safe exposure to psilocybin, as determined using clinical judgement of past and present medical and psychiatric history by any specialist psychiatrist or registered medical professional under the authorized delegation of a specialist psychiatrist.
2. First-degree relative with a diagnosed psychotic disorder.
3. Scores from the screening psychiatrist (or registered medical professional under the authorized delegation of a specialist psychiatrist) and baseline (S-STS) that indicate that the participant is of clinically significant risk of suicide. A decision will be formed based on S-STS scores and used in combination with other clinically significant data at screening. Sites should refer to the medical monitor if required.
4. Has attempted suicide in the twelve months preceding the screening visit.
5. Current (< 1 year) alcohol or drug misuse as identified as moderate or severe during screening in accordance with Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria, using the MINI 7.0.2, not able or willing to abstain from alcohol consumption in the period 12 hours prior to the dosing session.
6. Any other reason that might prevent a participant from engaging in therapeutic preparation and integration sessions.
7. Anyone who has taken a microdose of psilocybin within 5 days of baseline, taken a higher dose of psilocybin (e.g., dried mushrooms or capsules) within 30 days of baseline and experienced euphoria, hallucinations, or altered mental status, or used any classic psychedelics (LSD, ibogaine, ayahuasca, DMT, mescaline) within 3 months prior to baseline.

Medical Exclusion Criteria:

1. Diagnosed with brain metastases, glioblastoma, phaeochromocytoma, bowel obstruction or intestinal failure, active carcinoid syndrome, uncontrolled hypercalcaemia, or uncontrolled diabetes mellitus or insipidus.
2. Currently taking or planning to take any of the following: any typical or atypical antipsychotic and monoamine-oxidase inhibitors. Participants with prior use of these medications must be willing to discontinue their use for at least 2 weeks prior to the baseline visit and to Day 28.
3. Currently taking or planning to take any anticonvulsant or mood stabilizer, including carbamazepine, lithium, phenytoin, and valproate. Participants with prior use of these medications must be willing to discontinue their use for at least 1 week prior to the baseline visit and to Day 28.
4. Any form of fungal allergy.
5. Positive pregnancy test at screening, women who are breastfeeding or of childbearing potential who are unwilling or unable to use an effective form of contraception (or abstinence) for the study period and for 1 month post PEX010 dose will be excluded. Women will be required to conduct a serum pregnancy test at the in-person screening visit and urine test prior to dosing session. Male participants who do not agree to use contraception for the study period and for 90 days post PEX010 dose to mitigate the risk of pregnancy will also be excluded. Note: Refer to Section 4.3.2.1 for further details about contraception.
6. A diagnosis of epilepsy or at significant risk of seizures based on medical history.
7. Cardiovascular conditions including stroke and/or myocardial infarction (less than one year before providing informed consent), uncontrolled hypertension (blood pressure > 140/90 mmHg) or clinically significant arrhythmia at screening. Results are exempt if they are a direct result of the participant's cancer diagnosis and do not present a risk to administration of psilocybin, following discretion of the investigator.
8. Anyone who, at screening, has clinically significant findings on physical examination, including resting vital signs (HR below 40 or above 120 bpm, blood pressure below 90/60 or above 140/90), ECG (QTcF > 450 msec for males and >470 for females), and positive alcohol breath test. Note: Inclusion of individuals with any out-of-range values, including blood pressure, is at the discretion of the Investigator.
9. Liver dysfunction at screening as defined by AST and/or ALT > 1.5 times the upper level of normal or upper reference range. Results are exempt if they are a direct result of the participant's cancer diagnosis and do not present a risk to the administration of psilocybin, following discretion of the investigator.
10. Renal Function: estimated glomerular filtration rate <60 mL/min (calculated using Chronic Kidney Disease Epidemiology Collaboration) unless this is a direct result of the cancer diagnosis and does not present a risk to the administration of psilocybin, following the discretion of the investigator.
11. Any clinically significant laboratory abnormality(s) that in the opinion of the investigator would present a risk to the administration of psilocybin.
12. Any clinically significant renal, pulmonary, gastrointestinal, hepatic, or other illness that could affect the interpretation of results or be a potential health risk for the person if they were to be included in the study. Results are exempt if they are a direct result of the participant's cancer diagnosis and do not present a risk to administration of psilocybin, following discretion of the investigator.
13. Below 18 or above 32kg/m2 Body Mass Index (BMI) score at Screening.
14. Anyone with organic brain injury or diagnosed with any cognitive impairment.
15. Positive urine drug test for non-prescribed psychoactive substances at the dosing session visit. Positive urine drug test for psychoactive substances at the in-person screening should be referred to the medical monitor. Note: Testing may be repeated once at the discretion of the Investigator.
16. Anyone on a research study of an investigational drug or who has been on a clinical trial within 3 months of enrolment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-05-21 (Estimated); Study Completion 2026-08-21 (Estimated)

PRIMARY OUTCOMES:
Anxiety Severity | Comparison between treatment groups in the change from baseline in the Hamilton Anxiety Rating Scale (HAM-A) total score at Week 10 after a single PAP cycle.
  To assess the change in anxiety severity in participants with Adjustment Disorder (AjD) due to a cancer diagnosis, as measured by the Hamilton Anxiety Rating Scale (HAM-A). The Hamilton Anxiety Rating Scale (HAM-A) ranges from 0 to 56, with higher scores indicating greater anxiety severity.
Number of participants with treatment-related adverse events as assessed by CTCAE V5.0 | Assessment of Day 14 (dosing day) vital signs (pre-dose and prior to discharge).
  To assess the safety and tolerability of a single dose of PEX010 (25 mg, 10 mg and 1 mg [low-dose comparator]) in people with AjD with a cancer diagnosis.
Safety and Tolerability of a Single Dose of PEX010 using the Sheehan Suicide Tracking Scale (S-STS) | Assessment of suicidality using the Sheehan Suicide Tracking Scale (S-STS) at baseline, Day 13, Day 15, Weeks 4, 6, and 10, and 3 months post-final cycle.
  To assess the safety and tolerability of a single dose of PEX010 (25 mg, 10 mg, and 1 mg [low-dose comparator]) in people with Adjustment Disorder (AjD) due to a cancer diagnosis, using the Sheehan Suicide Tracking Scale (S-STS). The Sheehan Suicide Tracking Scale (S-STS) is a clinician-rated measure of suicidality that assesses suicidal ideation and behaviour. The scale consists of 14 items, with scores ranging from 0 to 60, where higher scores indicate greater suicidality risk.

CONTACTS AND LOCATIONS:
Overall Officials: Clive Ward-Able, Study Director — Psyence Biomedical
Locations (3):
- Australia (3):
  - Mind Medicine Australia Clinic, Abbotsford, Victoria
  - Paratus Clinical Research Melbourne, Northcote, Victoria
  - Empax Centre, Leederville, Western Australia

IPD SHARING:
Plan to Share IPD: No
Study-level documents, such as the Study Protocol, Statistical Analysis Plan, Informed Consent Form, Clinical Study Report, and Analytic Code, may not be shared at this time due to proprietary and confidential information. These documents contain data or methodologies that are critical to the sponsor's intellectual property and the integrity of ongoing or future analyses.